CLINICAL TRIAL: NCT05356052
Title: Expanded Access: Pulsed, Inhaled Nitric Oxide (iNO) for the Treatment of Patients With Serious Disease or Conditions Associated With Pulmonary Hypertension
Brief Title: Expanded Access for Patients With Pulmonary Hypertension Associated With Pulmonary Fibrosis
Status: Available | Type: Expanded Access
Sponsor: Bellerophon (Industry)
Responsible Party: Sponsor
Other Study IDs: PULSE-EAP-002
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Fibrosis; Pulmonary Hypertension
Keywords: PF; Pulmonary Fibrosis; Pulmonary Hypertension; PH; Inhaled Nitric Oxide; iNO; Long Term Oxygen Therapy; LTOT; Oxygen; INOpulse; pulsed inhaled nitric oxide; fILD; fibrotic interstitial lung disease; portable pulsed inhaled nitric oxide
MeSH Terms: conditions — Pulmonary Fibrosis; Hypertension, Pulmonary

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Combination Product: INOpulse — Patients will be treated by means of an INOpulse device using an INOpulse nasal cannula

SUMMARY:
An expanded access program that provides INOpulse treatment to patients with serious disease or conditions associated with pulmonary hypertension associated with pulmonary fibrosis who are not able to participate in the Sponsor's ongoing Phase 3 REBUILD clinical.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (and assent as appropriate) prior to the initiation of any study mandated procedures or assessments.
2. Subjects greater than 18 years of age at the time of consent to study participation.
3. Subjects with pulmonary hypertension associated with a disease or condition that are not eligible to participate in current ongoing clinical trials.
4. Subjects are willing and considered in the judgement of the Investigator able to use the INOpulse device continuously for up to 24 hours per day.
5. Female patients of childbearing potential must have a negative pre-treatment pregnancy test (serum or urine). All female patients should take adequate precaution to avoid pregnancy.
6. Subjects, in the opinion of the Investigator that would benefit from iNO treatment.

Exclusion Criteria:

1. Subjects who require treatment with riociguat.
2. Clinical contraindication to inhaled nitric oxide, as deemed by the Investigator.
3. Subjects who require concurrent Positive Airway Pressure (PAP) or Positive End Expiratory Pressure (PEEP).
4. Concurrent use of benzocaine, dapsone, nitrites and nitrates (amyl nitrite, isosorbide, nitroglycerin, nitroprusside), phenazopyridine. or primaquine.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, MD, Study Director — Bellerophon Therapeutics